CLINICAL TRIAL: NCT01376648
Title: Study on the Relationship Between the Thyroid Hormones and the Activity of Brown Adipose Tissue in Human
Brief Title: Thyroid Hormones Effect on Brown Adipose Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Yiming Li, Division of Endocrinology and Metabolism
Other Study IDs: KY2009-257
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2009-11

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — TSH, TT3, TT4, fT3, fT4, γT3,Norepinephrine,Blood-fat,FPG,Insulin,Leptin,Aadiponectin,Retinol-binding protein 4,Fatty acid binding protein 4,IL-6,TNF-α,CRP,Monocyte chemotactic protein 1
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Brown adipose tissue (BAT) is important in energy expenditure through thermogenesis although the regulatory factors are not well known in humans. There is evidence suggesting that the thyroid hormones affect BAT functions in lower mammals, but the effects of the thyroid hormones on BAT activity in humans are still unclear. The objective of this study was to investigate the effects of thyroid hormones on glucose metabolism of BAT and other organs in humans.

DETAILED DESCRIPTION:
Twenty consecutive patients with Graves'-caused hyperthyroidism who are newly diagnosed and untreated will be studied at the Endocrine Department of Huashan Hospital, Fudan University. All subjects are screened and examined by two senior investigators. Putative BAT activity is determined by the integrated 18F-fluorodeoxyglucose (18F-FDG) PET-CT. After the first PET scan, hyperthyroid patients will be treated with Methimazole following clinical guidelines. None of them uses beta adrenergic blockade. The initial dose of methimazole employed is 10mg thrice a day. During follow-up, the thyroid hormone levels (free triiodothyronine and free thyroxine) will be measured every twenty days. The PET-CT scans and assessments will be repeated when the symptoms have disappeared and the thyroid hormone levels return to normal range. Then the dose of methimazole will be adjusted accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and untreated hyperthyroid patients
* Informed consent was obtained

Exclusion Criteria:

* History of other endocrine diseases
* Useing beta adrenergic blockade
* Pregnant women
* Pacemaker implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty Graves' disease-caused hyperthyroid patients who were newly diagnosed and untreated were included. All hyperthyroid patients were treated with Methimazole and had been followed up until their symptoms disappeared and the thyroid hormone levels went back to normal range.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, Dr., Study Chair — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China